CLINICAL TRIAL: NCT02619383
Title: Hyperbaric Oxygen Can Improve Erectile Dysfunction and Induce Penile Angiogenesis
Brief Title: HBOT Application in Erectile Dysfunction
Acronym: HBOTED
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Dr. Shai Efrati, Assaf-Harofeh Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 42/13
Record Dates: First submitted 2015-11-29; First posted 2015-12-02 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Erectile Dysfunction; Hyperbaric Oxygen Therapy
Keywords: HBOT; hyperbaric oxygen; DCE; ED; erectile dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HBOT (Experimental): All patients were treated with 40 daily hyperbaric sessions, 5 days a week, in a multiplace hyperbaric chamber (HAUX-Life-Support GmbH). Each session consisted of 90 minutes of exposure to 100% oxygen at 2 ATA with 5 minutes air breaks every 30 minutes and 1 meter per minute compression and decompression.
  Interventions: Device: Hyperbaric oxygen therapy

INTERVENTIONS:
Device: Hyperbaric oxygen therapy — The treatment comprised 40 daily hyperbaric sessions, 5 days a week, in a multiplace hyperbaric chamber (HAUX-Life-Support GmbH). Each session consisted of 90 minutes of exposure to 100% oxygen at 2 ATA with 5 minutes air breaks every 30 minutes and 1 meter per minute compression and decompression.
  Other Names: HBOT

SUMMARY:
Recent studies have shown that hyperbaric oxygen therapy (HBOT) can induce angiogenesis and improve impaired organ function. HBOT was also recently suggested as a possible therapy for ED due to surgical injuries. However, the effect of HBOT on non-surgical related ED has not been investigated to date.

The objective in this study was to assess the effect of HBOT on patients with ED by means of sexual function questionnaires and novel imaging techniques.

DETAILED DESCRIPTION:
A prospective analysis of men, age 18 years or older, with a clinical diagnosis of erectile dysfunction, reporting decreased and weakened nocturnal penile tumescence of six months duration or longer.

Patients were treated at The treatment comprised 40 daily hyperbaric sessions, 5 days a week, in a multiplace hyperbaric chamber (HAUX-Life-Support GmbH). Each session consisted of 90 minutes of exposure to 100% oxygen at 2 ATA with 5 minutes air breaks every 30 minutes and 1 meter per minute compression and decompression.

Sexual function Efficacy of the treatment was assessed using the International Index of Erectile Function (IIEF) questionnaire which was filled by all patients at baseline and within 2 weeks of the last HBOT session. In addition, assessing efficacy was the global efficacy question (GEQ) ("Did the treatment improve your erections?"), with a response of yes or no.

Six patients underwent two MRI scans 1-2 weeks prior to and after HBOT. Imaging was conducted in using a 3Tesla system (MAGNETOM Skyra, Siemens Medical Solutions, , Germany). The MRI protocol included anatomic T1 and T2 sequences and DCE. The MRI DCE sequence parameters are detailed in supplementary section.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* clinical diagnosis of erectile dysfunction
* reporting decreased and weakened nocturnal penile tumescence of six months duration or longer

Exclusion Criteria:

* penile anatomical defects,
* any active or history of malignancy including prostate cancer
* spinal cord injury
* any major psychiatric disorder uncontrolled with treatment
* claustrophobia
* chronic lung disease
* chronic middle ear or sinus diseases.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-06; Primary Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Sexual function | 3 months
  Efficacy of the treatment was assessed using the International Index of Erectile Function (IIEF) questionnaire. Primary outcome was measured by questions 3 and 4 (Q3 and Q4). Question 3 asks 'Over the past four weeks, when you have attempted sexual intercourse how often were you able to penetrate (enter) your partner?'. Question 4 asks 'Over the past four weeks, during sexual intercourse, how often were you able to maintain your erection after you have penetrated your partner?'
Sexual function | 3 months
  global efficacy question (GEQ) ("Did the treatment improve your erections?"), with a response of yes or no.

SECONDARY OUTCOMES:
Imaging of penile perfusion | 3 months
  Imaging was conducted in using a 3Tesla system (MAGNETOM Skyra, Siemens Medical Solutions, , Germany). The MRI protocol included anatomic T1 and T2 sequences and DCE.
  K-trans calculations were performed in four specific axial sections located in each CC at the level of the penis base for better localization and reduced variability (Figure-1). Another control K-trans measurement was performed at the psoas muscle at the point in pass at the groin. The relative change in penile K-trans values (in %) was calculated as (post HBOT value - pre HBOT value) / pre HBOT value * 100.
  MRI includes Gadolinium contrast injection which has allergy related issues.
Adverse events | 3 months
  Rate of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf-Harofeh Medical Center, Ẕerifin, Israel